CLINICAL TRIAL: NCT04112953
Title: Intraoperative Transesophageal Echocardiography Assessment of Portal Vein Flow and Renal Resistive Index As a Predictor of Acute Kidney Injury After Cardiac Surgery: A Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: TEE PF/RRI AKI IRB19-0599
Record Dates: First submitted 2019-09-04; First posted 2019-10-02 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: AKI
Keywords: transesophagel echocardiography cardiac surgery kidney function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Upcoming cardiac surgery: Subjects in this group will have an upcoming cardiac surgery with the use of cardiopulmonary bypass and no pre-existing renal insufficiency or failure

SUMMARY:
The purpose of this study is to better understand if transesophageal echocardiography during cardiac surgery can predict problems with kidney function after cardiac surgery.

DETAILED DESCRIPTION:
Informed consent will be obtained prior to surgery. Preoperative demographic and baseline clinical data will be collected. We will assess the patient's risk of postoperative AKI using the validated Cleveland clinic score based on preoperative risk factors and calculate the European System Operative Score Risk Evaluation score (EuroSCORE II). After standard anesthesia induction and intubation, a TEE probe will be inserted by a cardiac anesthesiologist, who is certified in intraoperative echocardiography. We will use a standard ultrasound machine (EPIQ 7 Philips;Philips, Bothell, WA). Images of the right or left kidney along with Doppler flow and velocities will be obtained prior to cardiopulmonary bypass (CPB), after CPB, and after chest closure. Images of the portal vein with Doppler flow and velocity will be obtained prior to CPB, after CPB, and after chest closure. Vitals signs and hemodynamic data will be collected concurrently during these times. (See Data Sheet) Concurrent ECG will be obtained to identify the phases of the cardiac cycle. Mean arterial pressure (MAP) will be maintained within 20% of baseline MAP with bolus or continuous infusion of vasopressors (phenylephrine, norepinephrine, epinephrine, vasopressin, ephedrine). Cardiopulmonary bypass management will be standard, with target systemic blood flow of 2.4L/min/m2. Postoperative data will include urine output, serum creatinine, calculated GFR (using Modification of Diet in Renal Disease [MDRD] method) hospital and ICU length of stay, and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are patients >18 years old getting elective cardiac surgery with the use of cardiopulmonary bypass at the University of Chicago Medical Center.

Exclusion Criteria:

* Exclusion criteria are preexisting renal insufficiency/failure (glomerular filtration rate < 60 ml/min/1.73 m2 [stage 2 chronic kidney disease] or dialysis, renal vein thrombosis, renal artery stenosis, significant aortic regurgitation (moderate to severe aortic regurgitation on preoperative or intraoperative TEE), liver cirrhosis, portal vein thrombosis, preoperative intra-aortic counterpulsation balloon pump, emergency surgery, inability to obtain flow velocity waveforms of renal/portal vasculature on TEE, and kidney or liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be included who are scheduled for a standard of care cardiac surgery with the use of cardiopulmonary bypass at the University of Chicago Medical Center who meet the study's inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Portal vein pulsatility | intra-operative measurement
  Pulsed-wave Doppler measurement of portal vein flow and portal hypertension

SECONDARY OUTCOMES:
Renal resistance index | intra-operative measurement
  A sonographic index to assess for renal arterial disease measured via pulsed-wave Doppler
ICU length of stay | 30 days post-operation
  Length of ICU stay at any point for 30 days post-operation will be recorded
Hospital length of stay | 30 days post-operation
  Length of Hospital stay up to 30 days post-operation will be recorded
30-day mortality | 30 day post-operation
  Standard measure post

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared